CLINICAL TRIAL: NCT01482156
Title: An Open-label, Multi-center Phase I Dose-finding Study of RAD001 (Everolimus, Afinitor®) in Combination With BEZ235 in Patients With Advanced Solid Tumors
Brief Title: Dose Finding Study of RAD001 (Everolimus, Afinitor®) in Combination With BEZ235 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001X2109; 2011-001425-24 (EudraCT Number)
Record Dates: First submitted 2011-09-26; First posted 2011-11-30 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2015-11

CONDITIONS: Advanced Solid Tumors; Metastatic Breast Cancer; Metastatic Renal Cell Carcinoma
Keywords: Advanced solid tumors; Metastatic renal cell carcinoma (mRCC); ER+/HER2-Metastatic breast cancer (MBC); Dose finding study; mTOR; Pl3K; BEZ235; RAD001; Everolimus; Afinitor®; ER+/HER2- metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus; dactolisib

ARMS (1):
- RAD001 + BEZ235 (Experimental): Patients will receive first dose of RAD001 at 2.5mg/5mg/10 mg weekly or 2.5mg/5mg daily in combination of BEZ235 at 50 mg/100 mg/200 mg/300 mg/400 mg twice a day. In the initial cohort of the dose finding phase, patients will receive a single 2.5 mg dose of RAD001 on Cycle 1 Day 1 and the combination therapy of RAD001 2.5 mg/week and BEZ235 200 mg bid starting on Cycle 1 Day 8. Dose escalation phase: patients will start RAD001 and BEZ235 on Cycle 1 Day 1 with both study drugs being administered at the center. Dose expansion phase: the first 15 patients enrolled at selected sites will take RAD001 as monotherapy from Day 1 to Day 7 (for PK sampling). The combination therapy of RAD001 and BEZ235 will start on Day 8. All remaining patients will receive the combination therapy of RAD001 and BEZ235 starting on Cycle 1 Day 1.
  Interventions: Drug: RAD001 + BEZ235

INTERVENTIONS:
Drug: RAD001 + BEZ235 — RAD001 is formulated as tablets of 2.5 mg and 5 mg strength, blistered in units of 10 tablets (for oral use) each. Blisters should be opened only at the time of dministration as the drug is both hygroscopic and light-sensitive. RAD001 should be administered immediately after a meal with a large glass of water. BEZ235 is supplied as 50-mg, 200-mg, 300-mg and 400-mg sachets (for oral use). BEZ235 is packaged in aluminum foil bags. Bags are packaged in a box. Patients will receive RAD001 in combination with BEZ235.
  Other Names: Afinitor

SUMMARY:
Study has two parts:

1. Dose-finding: to determine the maximum tolerated dose (MTD) and to evaluate the safety and tolerability of RAD001 (everolimus , Afinitor®) in combination with BEZ235 in patients with advanced solid tumors.
2. Dose-expansion: to assess safety and tolerability of RAD001 and BEZ235 at the MTD in patients with ER+/HER2- metastatic breast cancer and metastatic renal cell cancer

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 years or older
* In the dose finding phase, patients with histologically or cytologically confirmed advanced solid malignancies that are metastatic or unresectable
* In the dose expansion phase, the enrollment will be limited to patients with:

Patients with metastatic renal cell carcinoma (mRCC) whose disease had progressed despite prior treatment with VEGFR-TKI (vascular endothelial growth factor receptor tyrosine kinase inhibitor) therapy (at least one but no more than two lines of VEGFR-TKI therapy) Patients with metastatic breast cancer (MBC) which is ER+/HER2-, whose disease had progressed despite prior treatment with at least one but no more than two lines of chemotherapy and at least one prior line of endocrine therapy in the metastatic setting

* WHO performance status of 0-2
* Lab parameters within specifically defined criteria
* Patients with measurable disease per RECIST 1.0

Exclusion Criteria:

* Patients who have previously received mTOR inhibitors or PI3K inhibitors
* Patients with CNS metastases unless previously treated with surgery, whole-brain radiation or stereotactic radiosurgery plus the disease having been stable for at least 2 months without steroid use for at least 1 month prior to the first dose of RAD001 and BEZ235. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs.
* Major surgery within 2 weeks prior to study enrollment
* Patient taking anti-cancer drug concomitantly
* Received radiation within 4 weeks prior to study enrollment (2 weeks if limited field radiation)
* Receive chemotherapy 4 weeks prior to study enrollment
* Received live attenuated vaccines within 1 week prior to study enrollment
* History of HIV
* Any other severe and/or uncontrolled medical condition

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Probability of a Dose Limiting Toxicity (DLT) by the end of the first treatment cycle (DLT) | First treatment cycle (28 days)
  The maximum tolerated dose (MTD) and the dose limiting toxicities during the first cycle of treatment
Incidence of DLT in patients by the end of the first treatment cycle in the co-administration of RAD001 and BEZ235 | First treatment cycle (28 days)
  Frequency of DLTs during the first cycle of treatment
Number of participants with adverse events and serious adverse events. | 12 months
  Measured by abnormal safety laboratory parameters, changes in electrocardiograms (ECGs), changes in vital signs and changes in physical examination parameters.

SECONDARY OUTCOMES:
Time versus blood concentration profiles | First treatment cycle ( 28 days)
  Analysis of pharmacokinetic parameters in blood samples
Overall Response Rate (ORR) (Complete Response (CR) + Partial Response (PR)) according to local assessments by RECIST 1.0 for renal cell carcinoma (RCC) and metastatic breast cancer (MBC) in dose expansion phase | 8 weeks
  CT or MRI imaging parameters to determine the overall response rate (complete response, partial response, stable disease, or progressive disease) according to the RECIST 1.0 criteria.
Progresive Free Survival (PFS) according to local assessments by RECIST 1.0 for renal cell carcinoma (RCC) and metastatic breast cancer (MBC) in dose expansion phase | 8 weeks
  CT or magnetic resonance imaging (MRI) imaging parameters to determine the PFS according to the RECIST 1.0 criteria
Duration of response (DoR) according to local assessments by RECIST 1.0 for RCC and MBC in dose expansion phase | 8 weeks
  CT or MRI imaging parameters to determine the duration of response according to the RECIST 1.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (3):
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - Washington University School of Medicine Washington University (16), St Louis, Missouri
  - Medical University of South Carolina SC, Charleston, South Carolina
- Novartis Investigative Site, Wilrijk, Belgium
- France (2):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Montellier Cedex 5
- Novartis Investigative Site, Verona, VR, Italy
- Novartis Investigative Site, Auckland, New Zealand
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, High Heaton, Newcastle Upon Tyne, United Kingdom

REFERENCES:
- See also: Results for CRAD001X2109 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14406